CLINICAL TRIAL: NCT00217932
Title: Double-Blind, Placebo-Controlled Study of Depakote (Divalproex Sodium) in Children With Temper Outbursts and Severe Mood Swings
Brief Title: Effectiveness of Divalproex Sodium (Depakote) in Treating Children With Temper Outbursts and Severe Mood Swings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00451-1; K02-00451-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2006-04

CONDITIONS: Mood Disorders
Keywords: Behavioral Disorders
MeSH Terms: conditions — Mood Disorders; Mental Disorders | interventions — Valproic Acid

INTERVENTIONS:
Drug: Divalproex Sodium (Depakote)

SUMMARY:
The purpose of this study is to determine the effectiveness of divalproex sodium (Depakote) versus placebo in treating children with temper outbursts and severe mood disorders.

DETAILED DESCRIPTION:
Depakote has been used to treat seizures in children for more than 20 years. The purpose of this study is to determine the effectiveness of divalproex sodium (Depakote) in treating children with temper outbursts and severe mood disorders.

This study will last 12 weeks. Participants will be randomly assigned to receive either 250 mg Depakote or placebo. The dose of medication will increase at the end of Week 1 to 500 mg of either depakote or placebo; participants will remain on this dose through Week 5. At Week 6, participants will cross-over and receive the other treatment (either depakote or placebo), which they will take through Week 12. Study visits will occur weekly and will include a physical exam, blood and urine tests, and self-reports of adverse events. In addition, caregivers will complete reports about mood swings throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Explosive Mood Disorder (EMD)
* Explosive temper as evidenced by four or more outbursts of rage, property destruction, or fighting per month
* Mood liability as evidenced by multiple, daily, distinct shifts from normal to irritable mood with withdrawn or boisterous behavior, occurring without a clear precipitant
* History of an EMD for one year without treatment
* EMD symptoms resulting in impairment in two or more of the following areas: school, the law, family, substance use, peers, or work
* EMD symptoms do not occur only during substance toxicity or withdrawal
* EMD symptoms are not confined to a single setting or context
* Parent and child willing to consent to study
* Inadequate response to an adequate trial (8 weeks) of psychotherapy and/or family therapy

Exclusion Criteria:

* Meets criteria for pervasive developmental disorder or childhood schizophrenia
* Seizure or other neurologic disturbance
* Pregnant
* Moderate to severe mental retardation
* Physical exam or laboratory results with significant abnormalities
* Positive Hepatitis screen test
* Liver dysfunction
* Active suicidal or homicidal ideation
* History of suicide attempts
* History of barbiturate use
* Unequivocal manic or hypomanic episode
* Meets criteria for attention deficit hyperactivity disorder (ADHD) and has not failed a trial of psychostimulants for ADHD
* Meets criteria for major depression in prepuberty
* If female, unwilling to use an effective method of contraception for the duration of the study
* Mitochondrial disease or family history of mitochondrial disease

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 2000-09; Study Completion 2005-08

PRIMARY OUTCOMES:
Reduction in symptoms of explosive mood disorder; measured throughout the study and at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Donovan, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States